Official Title: An Open-Label Evaluation of the Safety and Tolerability of SAGE-718 in

Participants with Mild Cognitive Impairment or Mild Dementia Due to

Alzheimer's Disease

NCT Number: NCT04602624

**Document Date:** SAP Version 1.0: 01 November 2021

# 9. STATISTICAL METHODS ANALYSIS PLAN

Statistical Analysis Plan (SAP) v1.0, 01 Nov 2021



Statistical Analysis Plan (SAP) v1.0 Version Date: 01-Nov-2021

> Sponsor: Sage Therapeutics Protocol no: 718-CNA-201

# Statistical Analysis Plan (SAP)

| Protocol Title: | An Open-Label Evaluation of the Safety and Tolerability of SAGE-718 in Participants with Mild Cognitive Impairment or Mild Dementia Due to Alzheimer's Disease |
|---|---|
| Protocol Version No./Date: | 2.0/23-Sep-2020 |
| CRF Version No./Date: | 1.0/07-Apr-2021 |
| SAP Version No./Date: | 1.0/01-Nov-2021 |

# 1.0 Approvals

| Sponsor | |
|---|---|
| Sponsor Name: | Sage Therapeutics, Inc. |
| Representative/ Title: | DocuSigned by: |
| Signature /Date: | Signer Name: Signing Reason: I approve this document Signing Time: 01-Nov-2021 11:34 EDT |
| Representative/ Title: | DocuSigned by: |
| Signature /Date: | Signer Name: Signing Rescrit approve this document Signing Time: 01-Nov-2021 11.49 EDT |
| PRA | |
| / Title: | |
| Signature /Date: | Signed by Reason Tam approving this document. Date & Time: 01 Nov 2021 08:44 AM -06:00 Document. |
| Biostatistician (Owner)<br>/ Title: | , Principal Biostatistician |
| Signature /Date: | Signed by: Principal Biostatistician Reason: I am approving this document. Date & Time: 01 Nov 2021 10:24 AM -04:00 |

(NOTE: Electronic Signatures should only be used if all parties have the ability to eSign.)



# 2.0 Change History

| Version/Date | Change Log |
|-------------------|----------------------------------|
| 0.1 / 28-Oct-2020 | Created as a new, Stable version |
| 1.0 / 01-Nov-2021 | Final Signed version |



# 3.0 Table of Contents

| | Approvals | |
|--------|---------------------------------------------------------|-----|
| | Change History | |
| 3.0 | Γable of Contents | 3 |
| | Purpose | |
| 5.0 \$ | Scope | 5 |
| 6.0 I | ntroduction | 5 |
| 6.1 ( | Changes from the Protocol | 5 |
| | Protocol Modifications | |
| | Modifications to the Approved Clinical Study Protocol | |
| 7.2 | Modifications to the Approved Statistical Analysis Plan | 6 |
| 7.3 [ | Modifications to the Approved DMC Charter | . 6 |
| 8.0 \$ | Study Objectives | 6 |
| 8.1 F | Primary Objective | . 6 |
| 909 | Study Endpoints | - 6 |
| | Primary Endpoint | |
| | Secondary Endpoints | |
| 0.2 | Secondary Endpoints | |
| 10.0 | Study Design | { |
| | Overall Design | |
| | Sample Size Considerations | |
| | Randomization | |
| | Analysis Sets. | |
| | Safety Set. | |
| 11.2 | Full Analysis Set | ` |
| 40.0 | Interine Analyses | Ţ, |
| | Interim Analyses | |
| | Statistical Methods | |
| | General Statistical Methodology | |
| | Participant Analysis Sets. | |
| 13.3 | Participant Disposition | 10 |
| 13.4 | Eligibility Criteria Violations and Protocol Deviations | 11 |
| | Demographic and Baseline Characteristics | |
| | Medical and Surgical History | |
| 13.7 | Physical/Neurological Examinations | 11 |
| | , -g | - |



| 13.8 Prior and Concomitant Medications | |
|---|---|
| 13.9 Treatments | |
| 13.9.1 Extent of Investigational Product Exposure and Treatment Adherence | 12 |
| 13.10 Visit Windows | 12 |
| 16.0 Safety and Tolerability Analyses | 30 |
| 16.1 Adverse Events | 30 |
| 16.1.1 Deaths and Serious Adverse Events (SAEs) | 30 |
| 16.2 Clinical Laboratory Evaluations | |
| 16.3 Physical/Neurological Examinations | 34 |
| 16.4 Vital Signs | |
| 16.5 12-Lead Electrocardiogram | |
| 16.6 Columbia-Suicide Severity Rating Scale (C-SSRS) | |
| 17.0 References | |
| 18.0 Glossary of Abbreviations | |
| 19.0 Appendix | |
| 19.1 Appendix-A Schedule of Study Assessment | |
| 19.2 Appendix-B Prior and Concomitant Medication Start/Stop Date Imputation | |
| 19.3 Appendix-C Adverse Event Start/Stop Date Imputation | |
| 19.4 Appendix-D Calculation of years since diagnosis of Alzheimer Disease | |
| The second of the second of th | |
| 10.6 Appendix E Tables Figures and Listings | 50 |



# 4.0 Purpose

The Statistical Analysis Plan (SAP) describes the statistical methods to be used during the reporting and analyses of data collected under Sage Therapeutics Protocol 718-CNA-201: An Open-Label Evaluation of the Safety and Tolerability of SAGE-718 in Participants with Mild Cognitive or Mild Dementia due to Alzheimer's Disease (AD).

# 5.0 Scope

This SAP describes the statistical methods to be used during the reporting and analyses of data collected from Sage Therapeutics Protocol 718-CNA-201, titled "An Open-Label Evaluation of the Safety and Tolerability of Sage-718-201 in Participants with Mild Cognitive or Mild Dementia due to AD

The Statistical Analysis Plan outlines the following:

- Study Objectives
- Study Design
- Study Endpoints
- The Analysis sets
- Applicable Study Definitions
- Statistical Methods

#### 6.0 Introduction

This is an open-label study evaluating the safety and tolerability of SAGE-718 s in participants with MCI or mild dementia due to AD. Eligible participants with a confirmed diagnosis of MCI or Mild dementia due to AD, according to the National Institute on Aging-Alzheimer's Association 2011 diagnostic guidelines, which will be confirmed via the CDR® Dementia Staging Instrument at screening will receive a 3.0 mg dose of SAGE-718 daily for 14 days.

This SAP should be read in conjunction with the study protocol and case report form (CRF). This version of the plan has been developed using the protocol Version 2, dated 23 September 2020 and CRF dated 07-Apr-2021.

Changes to the protocol will require an SAP amendment ONLY if the changes are to a principal feature of the protocol.

Final approval of the SAP by the Sponsor and PRA will occur prior to database lock. Any changes made to the SAP after the clinical database lock, along with the justification for the changes, will be described in the CSR.

# 6.1 Changes from the Protocol

- Protocol section 13.6.6 mentions the prior and concomitant medications will only be listed. Along
  with the listing a summary table will also be provided.
- Protocol section 13.4 mentions that Medical history will be only listed. Besides listing medical history will also be summarized.



 Alzheimer's disease history will be summarized and listed as per the data collected on the CRF page.



### 7.0 Protocol Modifications

7.1 Modifications to the Approved Clinical Study Protocol

Protocol version 2.0 is amended to revise the scheduled procedures and eligibility criteria to include more prospective participants.

- 7.2 Modifications to the Approved Statistical Analysis Plan This is the first version of SAP
- 7.3 Modifications to the Approved DMC Charter Not applicable

# 8.0 Study Objectives

- 8.1 Primary Objective
  - Evaluate the safety and tolerability of orally administered SAGE-718 in participants with mild cognitive impairment (MCI) or mild dementia due to Alzheimer's disease (AD).



# 9.0 Study Endpoints

- 9.1 Primary Endpoint
  - Incidence of treatment-emergent adverse events (TEAEs)



# 9.2 Secondary Endpoints

- Change from baseline in vital signs, clinical laboratory analytes, and electrocardiograms (ECGs).
- Change from baseline for responses on the Columbia

  Suicide Severity Rating Scale (C-SSRS).







# 10.0 Study Design

# 10.1 Overall Design

This study will enroll up to 22 participants that complete 14 days of dosing in this study. Additional participants may be dosed if the early discontinuation rate is >10%. Participants will be enrolled from approximately 5 sites in the US.

| This is an open-label study evaluating the safety and tolerability of SAGE-718 |
|---|
| in participants with MCI or mild dementia due to AD. Eligible participants |
| with a confirmed diagnosis of MCI or mild dementia due to AD, according to the National Institute on Aging- |
| Alzheimer's Association 2011 diagnostic guidelines, which will be confirmed via the CDR® Dementia |
| Staging Instrument will receive a 3.0 mg dose of SAGE-718 daily for 14 days within 1 hour of 30g fat meal. |

The study consists of a Screening Period, a Baseline Period, a Treatment Period, and a Follow-Up Period. The Screening Period begins with the informed consent process for prospective participants, including caregivers. Subsequent screening assessments will be performed between Day -21 and Day -8 to determine eligibility, including assessments of vital signs, clinical laboratory tests, electrocardiogram (ECG), magnetic resonance imaging (MRI) of the brain, and C-SSRS. An electroencephalogram (EEG) will also be performed preferably not in a fasting state.

<u>The Baseline Period</u> will occur from Day -7 through Day -1. During this period, each participant will receive dietary counseling to aid in choosing a morning meal containing approximately 30 g fat for dosing. On Day -7 (±1 day), participants will visit the clinic for confirmation of continued eligibility





and collection of baseline safety data. The Treatment Period will begin on Day 1 and continue through Day 14. During this time, participants will self-administer 3.0 mg SAGE-718 (as six 0.5-mg oral tablets), once per day in the morning within 1 hour after initiating a meal containing approximately 30 g of fat. Participants will continue in the clinic at scheduled visits and will track IP dosing and predose food intake in a participant diary. Participants will complete daily remote assessments Period clinic visits will occur on Day 1, Day 7 (±1 day), and Day 14. Following pre-dose procedures, participants will eat a morning meal and take the IP under staff supervision within 1 hour after initiating the meal. At scheduled clinic visits during the Treatment Period, safety, be performed, and study staff will dispense a sufficient amount of SAGE-718 for daily administration until the next scheduled study visit. In addition to weekly clinic visits, study staff will contact participants by telephone on Day 4 to document any TEAEs and/or changes in concomitant medications The Follow-Up Period, study staff will contact participants by telephone on Day 21 to document any TEAEs and/or changes in concomitant medications. Participants will then return to the clinic on Day 28 (±2 days) for a follow-up visit. No formal interim analysis or DSMB review are planned for this study. 10.2 Sample Size Considerations No formal sample size calculation was made for this study. Twenty participants completing 14 days of dosing are considered sufficient to assess preliminary safety and tolerability and for preliminary signalfinding after 14 days of repeated dosing with of SAGE-718. Assuming a 10% dropout rate, approximately 22 total participants will be required to obtain 20 completers. Additional participants may be dosed if the early discontinuation rate is >10%. 10.3 Randomization This study does not involve any randomization of participants. 11.0 Analysis Sets 11.1 Safety Set The Safety Set will include all participants who were administered at least one dose of investigational product (IP). Safety set will be used to describe the safety data.



# 12.0 Interim Analyses

There are no planned interim analyses for this study.

#### 13.0 Statistical Methods

### 13.1 General Statistical Methodology

All analyses will use SAS version 9.4 or higher.

Unless otherwise noted, continuous variables will be summarized using the number of observations (n), mean, standard deviation (std), median, first quartile (Q1), third quartile (Q3), minimum, and maximum values. The minimum and maximum values will be displayed to the same level of precision as the raw data; the mean, median, Q1, and Q3 values to one additional decimal place and the standard deviation to two additional decimal places.

Categorical variables will be summarized using counts and percentages. Percentages will be rounded to one decimal place, except 100% will be displayed without any decimal places, and percentages will not be displayed for zero counts.

All participants will be used in the analyses as per the analysis populations, using all non-missing data available. No imputation process will be used to estimate missing data.

For the purpose of all safety, and the last assessment prior to the first dose of study IP.

Prior and concomitant medication start/stop date imputation and adverse event start/stop date imputation are described in Appendix-B and Appendix-C, respectively.

AEs will be coded using Medical Dictionary for Regulatory Activities (MedDRA) version 23.1. All TEAEs are defined as an AE with onset after the first dose of IP.

#### 13.2 Participant Analysis Sets

The number and percentage of participants in the FAS, Safety, sets will be provided.

# 13.3 Participant Disposition

The number and percentage of participants screened, screen failed, enrolled in the study will be presented, together with the number and percentage of participants who discontinued from the study prematurely and a breakdown of the corresponding reasons for discontinuation as well as the number and percentage of participants who discontinued early from treatment and corresponding reasons.

Participant disposition will be summarized overall for the Safety analysis set, including the following:

- Number and percent of participants who completed the study
- Number and percent of participants who did not complete the study and reasons for early discontinuation of study

A by-participant disposition listing will be provided. In addition, a separate listing of screening failures with the primary reason for screen failures will be provided.



# 13.4 Eligibility Criteria Violations and Protocol Deviations

Protocol deviations identified during the study will be captured and categorized by the study team review as major and minor deviations on an ongoing basis. In addition, COVID-19 related protocol deviations such as remote telephone/video visit/assessment, home healthcare visit, missed visit/assessment, out of window visit/assessment, safety reporting, investigational product administration, and others will be documented and analyzed as appropriate.

A by-participant listing of all protocol deviations will be provided with columns identifying the following: date of the deviation, type of deviation (Major/Minor), deviation category, and verbatim description.

## 13.5 Demographic and Baseline Characteristics

Demographic and baseline characteristics, such as sex, race, age, height (cm), baseline weight (kg) body mass index (BMI) (kg/m²), and Clinical Dementia Rating (CDR) will be summarized using the Safety analysis set. Data will be summarized using descriptive statistics including sample size (n), mean, std, median, Q1, Q3, minimum, and maximum for continuous variables and numbers and percentages of participants for categorical variables.

Alzheimer's disease history will be summarized and listed by participants.

The baseline for weight, height and BMI is defined as the last non-missing value prior to the first dose of investigational product.

### 13.6 Medical and Surgical History

Medical/surgical history collected at screening will be coded using the Medical Dictionary for Regulatory Activities (MedDRA), Version 23.1. Medical/surgical history data will be summarized by system organ class (SOC) and preferred term (PT). A summary of medical/surgical history that is ongoing at the time of screening will be provided separately. Medical/surgical history will also be listed.

MRI results and amyloid-PET results will be listed by participants.

# 13.7 Physical/Neurological Examinations

A physical examination will be conducted at Screening (Day -21 to Day -8) and baseline (Day -7 and Day -1), as well as Days 14 and ET.

A full physical examination will occur at Screening and will include assessment of body systems (eg, head, eye, ear, nose and throat; heart; lungs; abdomen; and extremities) as well as neurological examination. Thereafter abbreviated physical examinations will include assessment of general appearance, cardiovascular, respiratory, gastrointestinal, and neurological systems, followed by a targeted physical examination as needed.

Clinically significant abnormalities found during Screening or during clinic visits will be reported on the medical history CRF; record clinically significant abnormalities or worsening conditions will be reported on the adverse event CRF, hence will be captured in AE displays. Therefore, no summaries will be provided for physical/neurological examinations.

#### 13.8 Prior and Concomitant Medications

The following analyses will use the Safety Set



All medications taken and procedures undergone during the study will be recorded.

Medications will be presented according to whether they are being taken prior to and/or during the study (concomitant). Prior medications are defined as those taken prior to the initiation of the start of the investigational product, and that ended prior to the IP. Concomitant medications are defined as those with a start date on or after the first dose of investigational product or those with a start date before the first dose of investigational product that is ongoing or with a stop date on or after the first dose of investigational product.

#### 13.9 Treatments

#### 13.9.1 Extent of Investigational Product Exposure and Treatment Adherence

The following analyses will use the Safety Set.

Total drug exposure (in mg) is defined as the total investigational product in mg for SAGE-718 that was taken during the study.

Total exposure duration to investigational product (in days) is defined as Date of last dose – date of first dose + 1. Note that this does not exclude days when the dose has been missed

Percent of the planned exposure received is defined as the total drug exposure, divided by planned exposure, times 100. For participants who complete the treatment period, planned exposure is 14 days of treatment planned times 3 mg. For participants who discontinued the treatment early, the planned exposure is the number of days (last date – first dose date + 1), times 3 mg.

Investigational product adherence (%) is defined as the number of tablets taken, divided by the number of tablets planned to be taken, times 100. The schedule of investigational product is six tablets per day. The number of tablets planned to be taken is defined as follows:

If the participant discontinues treatment within Day 2 and Day 14 (both inclusive), the number of tablets planned to be taken is the last dose day of investigational product × 6.

If the participant does not discontinue treatment, the number of tablets planned to be taken is 84 (6x14).

Investigational product exposure and adherence will be summarized descriptively and listed. The number and percentage of participants with investigational product adherence in categories(<80%, 80-100%, >100%) will be provided. Investigational product accountability will be listed.

All investigational product exposure data will be in by-participant listings, as well as a summary of treatment adherence.

#### 13.10 Visit Windows

The scheduled visits will not be windowed and will be used at a nominal visit value for analysis purposes. The unscheduled and early termination (ET) visit will be mapped to a scheduled visit for analysis. In order to accommodate as much data as possible into analysis, the windows in the table below have been widened compared to protocol-specified operational window, to have no gap between them; these windows are used for analysis purposes only. Once analysis visit windows are assigned, all visits, including scheduled visits, unscheduled visits, and ET visits will be eligible for being flagged as the "analyzed record" within the analysis window; a participant's individual analysis visit window could potentially contain more than 1 visit. In the event of multiple visits falling within an analysis window or in



case of a tie, the following rules will be used in sequence to determine the "analyzed record" for the analysis visit window:

- If the data from the scheduled visit is available, then the scheduled visit data will be used.
- If there is no data from the scheduled visit is available, the data closest to the scheduled study day for that window will be used.
- If there is a tie between the data in the number of days before and after the scheduled day, the later data will be used.

**Table 1: Visit Windows for Analysis** 

| Scheduled Visit<br>(+/1 window days) in protocol | Target Study Day | Study Day Window for Visit in Analysis |
|---|---|---|
| Day 1 | Day 1 (predose) | Day 1 (predose) or last non-<br>missing assessment before pre-<br>dose regardless of scheduled or<br>unscheduled visits |
| Day 7 (±1 day) | Day 7 | Day 2 - Day 10 |
| Day 14 (+1 day) | Day 14 | Day 11 - Day 17 |
| Day 28 / last dose + 14 days (±2 day) | Day 28 (last dose date<br>+ 14 days) | >= Day 26 (last dose date +12 days) |

Note: Parenthesized study day and study day window are for unscheduled visits, EOT and ET for participants who have discontinued treatment prematurely and such visit date is  $\geq 4$  days from the last dose of investigational product intake (ie, visit date – last dose date + 1 > 4).

The summary by visit will use the "analyzed records" only – at most one per participant. The data not flagged as the "analyzed record" will be included in listings. An unscheduled visit that does not fall under any analysis window will remain in the database and will be included in the listings.





















Sponsor: Sage Therapeutics





















Sponsor: Sage Therapeutics



























Sponsor: Sage Therapeutics





# 16.0 Safety and Tolerability Analyses

All safety analyses will be performed using the safety analysis set. Baseline for safety data is defined as the last non-missing value prior to the first dose of the investigational product.

Safety and tolerability of SAGE-718 will be evaluated by treatment-emergent adverse events (TEAEs) and change from baseline vital signs, clinical laboratory analytes, electrocardiograms (ECGs), safety electroencephalogram (EEG), and responses on the Columbia–Suicide Severity Rating Scale (C-SSRS). Safety data will be listed by the participant and summarized using descriptive statistics (mean, median, range, percentages).

#### 16.1 Adverse Events

TEAEs are defined as any AEs with an onset date on or after the date of the first dose of IP or any worsening of a preexisting medical condition/AE with onset after the start of IP and throughout the study. An AE leading to treatment discontinuation is defined as an AE with action taken of the investigational product as Drug Withdrawn. AEs will be coded using the Medical Dictionary for Regulatory Activities MedDRA version 23.1.

An overall summary of TEAEs, including the number of events, reported, the number and percentage of participants reporting at least one TEAE, the number and percentage of participants reporting at least one related TEAE, Number and percentage of participants by maximum severity, the number and percentage of participants discontinuing due to an adverse event, the number and percentage of participants with at least one serious adverse event, and the number and percentage of deaths will be presented.

A breakdown of the number and percentage of participants reporting each TEAEs, categorized by System Organ Class (SOC) and preferred term (PT), will be presented. Note that counting will be by a participant, not event, and participants are only counted once within each SOC and PT.

A further tabulation of these data, categorized by relationship (to SAGE-718), will be presented. Participants with multiple events within a particular body system or preferred term will be counted under the category of their drug-related event (related and not related) within SOC and PT. Relationship to SAGE-718 is categorized as related or not related.

A summary of events reported, categorized by severity, will also be provided. Participants with multiple events within a particular SOC and PT will be counted under the category of their most severe event in the following order: severe> moderate> mild within that SOC and PT.

A summary of adverse events leading to discontinuation of SAGE-718 will be provided, grouped by body system and preferred term.

All adverse events (including non-treatment-emergent events) recorded on the CRF will be listed.

Handling of missing AE start dates is defined in Appendix-C. Missing data for severity or relatedness to treatment will not be imputed.

#### 16.1.1 Deaths and Serious Adverse Events (SAEs)

All deaths and SAEs will be provided in by-participant listings.

### 16.2 Clinical Laboratory Evaluations

Laboratory assessments for biochemistry, coagulation, hematology, urinalysis, and serology, will be collected at screening, Day -1, Day 7, Day 14, and Day 28. The clinical laboratory tests to be performed for monitoring safety are listed in **Table 4**. Laboratory assessments will be summarized (n, mean, std,



median, Q1, Q3, minimum, and maximum) along with the change from baseline by each scheduled post-baseline visit. The International System of Unit (SI) will be used.

For the laboratory results that is "< or = x", where x is a number as collected in the data, the numeric part of the result will be used in the calculation in the summary tables. The same is true if the result is presented as below limit of quantification (BLQ) and a lower limit of quantification (LLOQ) value is provided – LLOQ value will be used for calculation in the summary tables. The actual results as collected will be displayed in the listings.

Summary tables on lab parameters will include descriptive statistics for the observed values and changes from baseline by scheduled assessment timepoint in hematology, serum chemistry, coagulation, and quantitative urinalysis test results.

**Table 4 Clinical Laboratory Tests** 

| Hematology | Serum Chemistry | Urinalysis | Coagulation |
|---|---|---|---|
| Hematology Red blood cell count Hemoglobin Hematocrit White blood cell count with differential Platelet count Red Blood Cell Indices (MCV, MCH, MCHC) Reflex to Red blood cell morphology if indices are abnormal | Serum Chemistry Alanine aminotransferase Albumin Alkaline phosphatase Aspartate aminotransferase Total bilirubin Direct bilirubin Indirect bilirubin Total protein Creatinine Blood urea nitrogen Creatine kinase Gamma-glutamyl transferase | Urinalysis pH Protein Glucose Red blood cell Nitrite Leukocyte esterase Ketones Bilirubin Urobilinogen | Coagulation Activated partial Thromboplastin time Prothrombin time International normalized ratio |
| apnormai | | Urobilinogen | |
| | Thyroid stimulating hormone (TSH) | | |

If a normal range is provided for the parameter, out-of-range values will be flagged as low or high, where applicable, in the participant data listings



The number and percentage of participants with potentially clinically significant (PCS) values will be provided in separate displays in hematology, serum chemistry, and liver function tests provided for such occurrence by time point.

PCS values will be identified for specific laboratory parameters as outlined in Table 5.

Liver function tests will be monitored closely for PCS values, and will be summarized for occurrence any time post-baseline for the following parameters for these PCS thresholds (for conditions involving more than one parameter, the results need to be from the same timepoint):

Alanine Aminotransferase: >3xULN, >5xULN, >10xULN Aspartate Aminotransferase: >3xULN, >5xULN, >10xULN

Alanine Aminotransferase or Aspartate Aminotransferase: >3xULN, >5xULN, >10xULN

Alkaline Phosphatase: >1.5xULN, >2xULN

Total Bilirubin: >1.5xULN, >2xULN

Total Bilirubin > 2xULN **AND** (Alanine Aminotransferase or Aspartate Aminotransferase >3xULN)
Total Bilirubin >2xULN **AND** Alkaline Phosphatase >2xULN **AND** (Alanine Aminotransferase or

Aspartate Aminotransferase >3xULN)

Any lab results considered clinically significant by the investigator will be captured as adverse events, hence will show up in AE displays.

Pregnancy test results will be listed but not summarized.

Table 5 Potentially Clinically Significant Values for Specific Laboratory Parameters

| Laboratory<br>Parameter | Gender | Units | Criteria for PCS Values (Observed values) | |
|---|---|---|---|---|
| | | | High | Low |
| Hematology | | | | |
| Hemoglobin | Male | g/L | >185 | <115 |
| | Female | g/L | >170 | <100 |
| Hematocrit | Male | Fraction of 1 | >0.55 | <0.385 |
| | Female | Fraction of 1 | >0.49 | <0.345 |
| Platelet count | | 10^9/L | >600 | <125 |
| White blood cell | | 10^9/L | >15 | <2.5 |
| Basophils | | 10^9/L | >0.5 | NA |
| Eosinophils | | 10^9/L | >1.5 | NA |
| Neutrophils | | 10^9/L | NA | <1.5 |
| Lymphocytes | | 10^9/L | >6.0 | <0.5 |
| Monocytes | | 10^9/L | >1.4 | NA |



| Laboratory<br>Parameter | Gender | Units | Criteria for PCS V | Criteria for PCS Values (Observed values) |
|---|---|---|---|---|
| | | | High | Low |
| Serum Chemistry | | | | |
| Albumin | | g/L | >70 | <28 |
| Blood urea nitrogen | | mmol/L | >10.71 | NA |
| Calcium | | mmol/L | >2.75 | <2.0 |
| Chloride | | mmol/L | >120 | <90 |
| Creatinine | | mmol/L | >3xULN or >3x<br>Baseline | |
| Gamma Glutamyl<br>Transferase | | | >3xULN | |
| Glucose | | mmol/L | >13.9 | <2.8 |
| Sodium | | mmol/L | >150 | <132 |
| Potassium | | mmol/L | >5.4 | <3.3 |
| Protein | | g/L | | <45 |
| Bicarbonate | | mmol/L | >34 | <18 |
| | | mmol/L | >120 | <90 |
| Phosphorus | | mmol/L | >1.94 | <0.61 |
| Liver Function Tests (LFT) | | | | |
| Bilirubin | | μmol/L | >2xULN | NA |
| Aspartate<br>Aminotransferase | | U/L | >3xULN | NA |
| Alanine<br>Aminotransferase | | U/L | >3xULN | NA |
| Alkaline Phosphatase | | U/L | >1.5xULN | NA |



# 16.3 Physical/Neurological Examinations

The occurrence of a physical examination, Neurological examination (yes/no), and the date performed will be listed by the participant.

### 16.4 Vital Signs

Vitals for the following parameters - respiratory rate (breaths/minute), oral temperature (degrees C), supine heart rate (beats/minute), supine systolic blood pressure (mmHg), supine diastolic blood pressure (mmHg), standing heart rate (beats/minute), standing systolic blood pressure (mmHg), standing diastolic blood pressure (mmHg), – are collected at Screening and on Days -7, -1, 1, 7, 14, and 28. Descriptive summaries of observed values and changes from baseline will be provided for vital sign parameters - by scheduled assessment time point. Additionally, the number and percentage of participants with PCS and potentially clinically significant change (PCSC) values will be summarized for such occurrence any time post-baseline. Potentially clinically significant values will be identified for vital sign parameters as outlined in Table 6.

Table 6 Potentially Clinically Significant Values and Change for Vital Sign Parameters

| Vital Sign | Units | Criteria for PCS Values<br>(Observed values) | | Criteria for PCSC values<br>(Change from Baseline<br>values) | |
|---|---|---|---|---|---|
| | | High | Low | Increase | Decrease |
| Heart rate (supine and standing) | Beats/min | >120 | <40 | NA | NA |
| Systolic Blood Pressure (supine and standing) | mmHg | >180 | <90 | ≥30 | ≥30 |
| Diastolic Blood pressure (supine and standing) | mmHg | >110 | <50 | ≥20 | ≥20 |
| Supine - Standing Systolic<br>Blood Pressure | mmHg | ≥20 | | | |
| Supine – Standing Diastolic<br>Blood Pressure | mmHg | ≥10 | | | |
| Orthostatic hypotension:<br>supine – standing SBP and<br>DBP | mmHg | SBP ≥20<br>and DBP<br>≥10 | | | |
| Possible Orthostatic<br>hypotension: supine –<br>standing SBP and DBP | mmHg | SBP ≥20 or<br>DBP<br>≥10 | | | |

The orthostatic vital sign - the change from supine to standing (Supine – Standing) in heart rate, systolic and diastolic blood pressure – will be summarized by scheduled assessment timepoint, at 1 and 3 minutes.


Any vital signs result considered clinically significant by the investigator will be captured as adverse events, hence will show up in AE displays. All vital sign assessments along with PCS will be listed in the listing.

### 16.5 12-Lead Electrocardiogram

Supine 12-lead ECGs will be performed in triplicate, and are collected on screening, days -1, 1, 7, 14, and 28. The following ECG parameters will be listed for each participant: heart rate (beats per minute), PR (msec), QRS (msec), QT (msec), and QTcF (msec).

The average of the triplicate values will be used in the summary, including baseline ECG values. The observed value at each time point and change from baseline at each post-baseline scheduled time point will be summarized. Each ECG is evaluated as 'normal', 'abnormal, not clinically significant' and 'abnormal, clinically significant'; the number and percentage of participants with at least one of the triplicate values in the categories of 'abnormal, clinically significant' and 'abnormal, not clinically significant' will be provided at baseline and each post-baseline scheduled assessment time point.

The number and percentage of participants with PCS and PCSC values will be summarized for such occurrence any time post-baseline. Potentially clinically significant values will be identified for ECG parameters as outlined in Table 7. A listing of ECG and QTcF PCS values will be provided.

Table 7 Potentially Clinically Significant Values and Change for ECG Parameters

| ECG | Units | Criteria for PCS Values (Observed val | Criteria for PC<br>(Change from | | |
|---|---|---|---|---|---|
| | | High | Low | Increase | Decrease |
| QTcF<br>Interval | msec | >450 but <=480<br>>480 but <=500<br>>500 | NA | >=30 to 60<br>>60 | NA |

### 16.6 Columbia-Suicide Severity Rating Scale (C-SSRS)

Suicidality will be monitored during the study using the C-SSRS. The C-SSRS is a questionnaire used to measure the presence and intensity of suicidal ideation and behavior. The C-SSRS will be completed at Screening, Days -7, -1, 1, 7, 14, and 28. The "Baseline/Screening" C-SSRS form will be completed at screening (lifetime history and past 24 months). The "Since Last Visit" C-SSRS form will be completed at subsequent time points.

Suicidal behavior and suicidal ideation will be summarized by visit for the Safety analysis set. The proportion of participants who meet the criterion for each of these categories at any post-baseline visit will be summarized as described in Table 8.



#### Table 8 C-SSRS Categories for Analysis

| Category | C-SSRS Item response is "YES" |
|---|---|
| Suicidal ideation | <ul> <li>Wish to be dead</li> <li>Non-specific active suicidal thoughts</li> <li>Active Suicidal Ideation with Any Methods</li> <li>Active Suicidal Ideation with Some Intent</li> <li>Active Suicidal Ideation with Specific Plan</li> </ul> |
| Suicidal behavior | <ul> <li>Preparatory Acts or Behaviour</li> <li>Aborted Attempt</li> <li>Interrupted Attempt</li> <li>Actual Attempt(non-fatal)</li> <li>Completed suicide [1]</li> </ul> |
| Suicidal Ideation or Behavior | Participant Engaged in Non-Suicidal Self-Injurious Behavior |

<sup>[1]</sup> Completed suicide is not collected at the screening visit.



#### 17.0 References

- ICH Harmonized Tripartite Guideline. Statistical Principles for Clinical Trials E9. International
  conference on harmonization of technical requirements for registration of pharmaceuticals for
  human use. 05 February 1998.
  <a href="http://www.ich.org/fileadmin/Public Web Site/ICH Products/Guidelines/Efficacy/E9/Step4/E9">http://www.ich.org/fileadmin/Public Web Site/ICH Products/Guidelines/Efficacy/E9/Step4/E9</a>
  Guideline.pdf
- ICH Harmonized Tripartite Guideline. Structure and Content of Clinical Study Reports E3. International conference on harmonization of technical requirements for registration of pharmaceuticals for human use. 30 November 1995. <a href="http://www.ich.org/fileadmin/Public Web Site/ICH Products/Guidelines/Efficacy/E3/E3 Guideline.pdf">http://www.ich.org/fileadmin/Public Web Site/ICH Products/Guidelines/Efficacy/E3/E3 Guideline.pdf</a>
- SAS/STAT 14.2 User's Guide, The Mixed Procedure. SAS Institute, Cary NC, 2016, pp. 6138-6275.
- SAS Programming to Calculate AUC in Pharmacokinetic Studies Comparison of Four Methods in Concentration Data. J. He. 2008. https://www.lexjansen.com/pharmasug/2008/sp/SP06.pdf



# 18.0 Glossary of Abbreviations

| Glossary of Abbrevia | ations: |
|---|---|
| AD | Alzheimer's Disease |
| AE | Adverse event |
| ATC | Anatomic Therapeutic Chemical |
| AUC <sub>0-t</sub> | Area under the plasma concentration-time curve, from time 0 to time t |
| AUC <sub>0-last</sub> | Area under the curve from the time of dosing to the time of the last measurable (positive) concentration |
| BLQ | Below the Limit of Quantification |
| CI | Confidence Interval |
| CV | Coefficient of Variation |
| C <sub>max</sub> | Maximum observed concentration. |
| COVID-19 | Coronavirus Disease 2019 |
| CRF | Case Report Form |
| CSR | Clinical Study Report |
| ECG | Electrocardiogram |
| eCRF | Electronic Case Report Form |
| IP | Investigational Product |
| LLOQ | Lower Limit of Quantification |
| MedDRA | Medical Dictionary for Regulatory Activities |
| PCS | Potentially Clinically Significant |
| PT | MedDRA Preferred Term |
| Q1 | First Quartile |
| Q3 | Third Quartile |
| SAP | Statistical Analysis Plan |
| SAE | Serious Treatment-emergent Adverse Event |
| SI | International System of Units |
| SOC | MedDRA System Organ Class |
| Std | Standard Deviation |
| TEAE | Treatment Emergent Adverse Event |
| WHO | World health Organization |



## 19.0 Appendix

## 19.1 Appendix-A Schedule of Study Assessment

| Study Period | Screening | Base | eline | | Trea | tment | | Follo | w Up |
|---|---|---|---|---|---|---|---|---|---|
| Study Day | D -21 to<br>D -8 | D -7<br>(±1 d) | D -1 | D 1 | D 4 a | | | D 21 a (±1 d) | |
| Informed consent b | X | | | | | | | | |
| Inclusion/exclusion criteria | X | X | X | | | | | | |
| Medical history and demographics c | X | | | | | | | | |
| Body weight | X | | | X | | X | X | | X |
| Body height | X | | | | | | | | |
| CDR | X | | | | | | | | |
| Test of Premorbid Functioning | X | | | | | | | | |
| Vital signs <sup>d</sup> | X | X | X | X | | X | X | | X |
| Physical examination <sup>e</sup> | X | X | X | | | | X | | |
| EEG <sup>f</sup> | X | | | | | | | | |
| 12-lead ECG g | X | | X | X | | X | X | | X |
| C-SSRS h | X | X | X | X | | X | X | | X |
| Clinical laboratory tests i | X | | X | | | X | X | | X |
| Alcohol test j | X | X | | | | | | | |
| Urine drug test | X | X | X | X | | X | X | | |
| FSH test k | X | | | | | | | | |
| Pregnancy test 1 | X | | X | | | | X | | X |
| Serology test <sup>m</sup> | X | | | | | | | | |
| MRI <sup>n</sup> | X | | | | | | | | |
| Study Period | Screening | Base | eline | | Trea | tment | | Follow | Up |



| Study Day | D -21 to<br>D -8 | D -7<br>(±1 d) | D -1 | D 1 | D 4 a | | D 14<br>or ET | D 21 a (±1 d) |
|---|---|---|---|---|---|---|---|---|
| Participant training p, q | | X | X | | | | | |
| Pamata assassments V | | | | | | | | |
| Remote assessments v | | | | | X (ana | - d-:1) | | |
| IP self-administration w | | | | | X (one | e daily) | ) | |
| IP dispensation <sup>x</sup> IP accountability <sup>y</sup> | | | | X | 2 | X | | |
| Safety telephone call | | | | | X | | | X |
| TEAEs/SAEs | | | | | X | | | |
| Concomitant medications <sup>z</sup> | | | | | X | | | |

Abbreviations: CDR = Clinical Dementia Rating Dementia Staging Instrument®; C-SSRS = Columbia—Suicide Severity Rating Scale; d = days; ECG = electrocardiogram; EEG = electrocarcephalogram; ET = early termination; FSH = follicle stimulating hormone; HIV = human immunodeficiency virus; IP = investigational product; MRI = magnetic resonance imaging; PET = positron emission tomography; SAE = serious adverse event; TEAE = treatment-emergent adverse event

Notes: In the event of ET, efforts should be made to collect the Day 14 visit assessments.

When scheduled for the same time point, procedures should be performed in the following order: vital signs, ECG, blood draws, morning meal, IP dosing, then any scheduled postdose assessments.

In the setting of public health advisories due to COVID-19, assessments scheduled to be conducted at the study site may be performed via telephone/video if feasible. For assessments that cannot be conducted by phone or video, an in-home visit may be conducted. Information about COVID-19 diagnosis, treatment, and quarantine status will be collected with the medical history, AEs, and prior and concomitant medications.

a Day 4 and Day 21 visits will occur via scheduled telephone calls.



Protocol no: 718-CNA-201 b Both study partners and participants are to be consented during the Screening Period. c In addition to full medical history, all nonpharmacological methods (eg. used to treat or prevent of AD are to be recorded. d Vital signs to include temperature, respiratory rate, heart rate, and blood pressure. Heart rate and blood pressure to be collected in supine position and standing position at all scheduled time points. When scheduled for the same visit, vital signs are to be assessed prior to ECG and blood collection. e Full physical examination to be conducted at Screening, abbreviated examinations thereafter. Unscheduled, symptom-directed physical examinations may also be conducted at the investigator's f EEG to be performed for all participants during Screening. If clinical events suspicious for seizure occur, an unscheduled 1-hour EEG will be performed (with a second follow-up 1-hour EEG at the discretion of the investigator). g ECG will be measured after the participant has been in the supine position for at least 5 minutes. h "Baseline/Screening" C-SSRS form at Screening and "Since Last Visit" C-SSRS form thereafter. i Samples for clinical laboratory assessments for hematology, biochemistry, coagulation, urinalysis, and serology to be collected ≤2 hours prior to dosing during the Treatment Period, and any time of day at other time points. Participants are to be in a fasted state for screening assessments only. j Alcohol testing will be performed in the clinic, either by urine dipstick or breathalyzer. k To confirm self-reported postmenopausal status in women only. I Serum pregnancy tests for all female participants at Screening; urine pregnancy tests will be conducted for all female participants who are not postmenopausal or surgically sterile at other scheduled time points. m To include testing for hepatitis B and C, HIV-1, and HIV-2 n Only in participants without an MRI report obtained within the 2 years preceding the Baseline Period p Where participant informed consent is given, samples for exploratory biochemical research and genetic testing will be collected after the collection of samples, according to the schedule in Table 3. q Participants and study partners will be trained to use all study-related software and devices. Additional guidance will be provided on choosing a meal with approximately 30 g of fat.



v Daily reminders will be sent to participants to complete assessments of

or in the clinic during the

Treatment Period (with observation by study staff during scheduled clinic visits).

- w On visit days during the Treatment Period, participants will self-administer IP in the clinic under the supervision of study staff after the predose assessments and consumption of a morning meal.
- x Study staff will dispense sufficient IP for daily dosing at home until the next scheduled visit. On Days 7 and 14, participants will return used IP packaging and any unused IP for site staff to document.
- y On Days 7 and 14, participants will return used IP packaging and any unused IP for site staff to document.
- z At Screening, include all psychotropic medications used within 12 weeks of informed consent, any other medications and supplements taken within 60 days of informed consent, and all medication used to treat AD, regardless of timing. After Screening, all changes to any medication or supplements should be captured.



## 19.2 Appendix-B Prior and Concomitant Medication Start/Stop Date Imputation

Imputation Rules for Partial Dates (D = day, M = month, Y = year)

| Parameter | Missing | Additional Conditions | Imputation |
|---|---|---|---|
| Start date for con meds | D only | M and Y same as M and Y of investigational product administration | Date of investigational product administration |
| | | M and/or Y not same as date investigational product administration | First day of month |
| | M and D | Y same as Y of investigational product administration | Date of investigational product administration |
| | | Y not same as Y of investigational product administration | Use Jan 01 of Y |
| | M, D, and Y | None - date completely missing | Day prior to date investigational product administration |
| Stop date for con meds | D only | M and Y same as M and Y of investigational product administration | Date of investigational product administration |
| | | M and/or Y not same as date of investigational product administration | Last day of month |
| | M and D | Y same as Y of investigational product administration | Date of investigational product administration |
| | | Y not same as Y of investigational product administration | Use Dec 31 |
| | M, D, and Y | None - date completely missing and NOT ongoing | Date of investigational product administration |

### 19.3 Appendix-C Adverse Event Start/Stop Date Imputation

| Parameter | Missing | Additional Conditions | Imputation |
|---|---|---|---|
| Start date for AEs | D | M and Y same as M and Y of investigational product administration | Date of investigational product administration |
| | | M and/or Y not same as date investigational product administration | First day of month |
| | D and M | Y same as Y of investigational product administration | Date of investigational product administration |
| | | Y prior to Y of investigational product administration but same as Y of screening date | Date of screening date |
| | D, M, Y | None - date completely missing | Date of investigational product |
| Stop date for AEs | D | M and Y same as M and Y of investigational product administration | Date of investigational product administration |
| | | M and/or Y not same as date of investigational product administration | Use last day of month |
| | D and M | Y same as Y of investigational product administration | Date of investigational product |
| | | Y not same as Y of investigational product administration | Use Dec 31 |
| | D, M, Y | None - date completely missing | No imputation, but assume ongoing |

Note: In all cases, if an estimated start date is after a complete stop date, use the first day of the stop date month. Similarly, if the estimated stop date is before a complete or imputed start date, use the last day of the start day month.



## 19.4 Appendix-D Calculation of years since diagnosis of Alzheimer Disease

| Observed | Missing | Formula to Calculate Duration |
|---|---|---|
| D,M,Y | | (Date of Enrollment – Date of Diagnosis + 1)/365.25 |
| M and Y | D | [Year (Date of Enrollment) – Year (Date of Diagnosis)] + [Month (Date of Enrollment) – Month (Date of Diagnosis)]/12 |
| Υ | D and M | [Year (Date of Enrollment) – Year (Date of Diagnosis)] |

Note: The number of years from the date of diagnosis to the date of enrollment, which will be derived based on the table above. No imputation will be done for missing diagnosis date (Year, Month, Day).

































# 19.6 Appendix-F Tables, Figures, and Listings

Table Number Title Population

| Table 14.1.1.1 | Subject Analysis Sets | All Screened Subjects |
|---|---|---|
| Table 14.1.1.2 | Subject Disposition | Safety Analysis Set |
| Table 14.1.1.3 | Major Protocol Deviations | Full Analysis Set |
| Table 14.1.2.1 | Demographic Characteristics | Safety Analysis Set |
| Table 14.1.3 | Prior Medications by ATC Classification and WHO Drug Dictionary Preferred Term | Safety Analysis Set |
| Table 14.1.4 | Concomitant Medications by ATC Classification and WHO Drug Dictionary Preferred Term | Safety Analysis Set |
| Table 14.1.5 | Medical and Procedures by System Organ Class and Preferred Term | Safety Analysis Set |
| Table 14.1.6 | Medical and Surgical History that are Ongoing at the time of Screening by WHO Drug Dictionary Preferred Term | Safety Analysis Set |
| Table 14.1.7 | Alzheimer Disease History | Safety Analysis Set |
| Table 14.1.8 | Summary of Exposure and Adherence | Safety Analysis Set |









| Table 14.3.1.1 | Overall Summary of Treatment-Emergent Adverse Events | Safety Analysis Set |
|---|---|---|
| Table 14.3.1.2 | Treatment-Emergent Adverse Events by System Organ Class and Preferred Term | Safety Analysis Set |
| Table 14.3.1.3 | Treatment-Emergent Adverse Events Leading to Discontinuation of the Study by System Organ Class and Preferred Term | Safety Analysis Set |
| Table 14.3.1.4 | Treatment-Emergent Adverse Events Leading to Interruption of Study treatment | Safety Analysis Set |
| Table 14.3.1.5 | Treatment-Emergent Serious Adverse Events by System Organ Class and Preferred Term | Safety Analysis Set |
| Table 14.3.1.6 | Treatment-Emergent Adverse Events with Outcome of Death by System Organ Class and Preferred Term | Safety Analysis Set |
| Table 14.3.1.7 | Treatment-Emergent Adverse Events Leading to Discontinuation of Study Treatment by System Organ Class and Preferred Term | Safety Analysis Set |
| Table 14.3.1.8 | Treatment-Emergent Adverse Events by System Organ Class, Preferred Term, and Relationship to IP | Safety Analysis Set |
| Table 14.3.1.9 | Treatment-Emergent Adverse Events by System Organ Class, Preferred Term, and Maximum Severity | Safety Analysis Set |



| | 1100 | DC01110. 7 10-CNA-201 |
|---|---|---|
| Table 14.3.3.1.1 | Hematology and Coagulation Results by Time Point | Safety Analysis Set |
| Table 14.3.3.1.2 | Potentially Clinically Important Postbaseline Hematology Results by Time Point | Safety Analysis Set |
| Table 14.3.3.2.1 | Biochemistry Results by Time Point | Safety Analysis Set |
| Table 14.3.3.2.2 | Potentially Clinically Important Postbaseline Biochemistry Results | Safety Analysis Set |
| Table 14.3.3.3.1 | Urinalysis Results by Time Point Part 1 Continuous ∀ariables | Safety Analysis Set |
| Table 14.3.3.3.2 | Urinalysis Results by Time Point Part 2 Categorical ∀ariables | Safety Analysis Set |
| Table 14.3.4.1 | Vital Sign Results by Time Point | Safety Analysis Set |
| Table 14.3.4.2 | Potentially Clinically Important Vital Sign Results | Safety Analysis Set |
| Table 14.3.5.1 | Electrocardiogram Results | Safety Analysis Set |
| Table 14.3.5.2 | Electrocardiogram Interpretations by Time Point | Safety Analysis Set |
| Table 14.3.5.3 | Potentially Clinically Important Electrocardiogram Results | Safety Analysis Set |
| Table 14.3.6 | Summary of Columbia–Suicide Severity Rating Scale (C-SSRS) Suicidal Ideation and Suicidal Behavior | Safety Analysis Set |



| Listing 16.1.7 Subject Enrollment Listing 16.2.1.1 Discontinued Subjects from Study Listing 16.2.1.2 Completion / Discontinuation of Investigational Product (IP) Listing 16.2.2 Protocol Deviations Listing 16.2.3.1 Subject Analysis Sets Listing 16.2.4.1 Demographic and Baseline Data All Screened Subjects Safety Analysis Set All Enrolled Subjects Listing 16.2.3.1 Demographic and Baseline Data Safety Analysis Set | | <u> </u> | 1010C01110. 7 10-CNA-201 |
|---|---|---|---|
| Listing 16.2.1.1 Discontinued Subjects from Study Safety Analysis Set Listing 16.2.1.2 Completion / Discontinuation of Investigational Product (IP) Safety Analysis Set Listing 16.2.2 Protocol Deviations Safety Analysis Set Listing 16.2.3.1 Subject Analysis Sets All Enrolled Subjects | | | |
| Listing 16.2.1.2 Completion / Discontinuation of Investigational Product (IP) Safety Analysis Set Listing 16.2.2 Protocol Deviations Safety Analysis Set Listing 16.2.3.1 Subject Analysis Sets All Enrolled Subjects | | | |
| Listing 16.2.2 Protocol Deviations Safety Analysis Set Listing 16.2.3.1 Subject Analysis Sets All Enrolled Subjects | | | |
| Listing 16.2.3.1 Subject Analysis Sets All Enrolled Subjects | Listing 16.2.1.2 | Completion / Discontinuation of Investigational Product (IP) | Safety Analysis Set |
| | Listing 16.2.2 | Protocol Deviations | Safety Analysis Set |
| Listing 16.2.4.1 Demographic and Baseline Data Safety Analysis Set | Listing 16.2.3.1 | Subject Analysis Sets | All Enrolled Subjects |
| | Listing 16.2.4.1 | Demographic and Baseline Data | Safety Analysis Set |



| Listing 16.2.4.2 | General Medical History | Safety Analysis Set |
|---|---|---|
| Listing 16.2.4.3 | Prior and Concomitant Medications | Safety Analysis Set |
| Listing 16.2.4.4 | Prior and Concomitant Procedures | Safety Analysis Set |
| Listing 16.2.5.1 | Administration of Investigational Product (Oral) | Safety Analysis Set |
| Listing 16.2.5.2 | Drug Accountability | Safety Analysis Set |
| Listing 16.2.5.3 | Treatment Adherence | Safety Analysis Set |

| Listing 16.2.7.1 | Adverse Events | Safety Analysis Set |
|---|---|---|
| Listing 16.2.7.2 | Subjects with Adverse Events with Outcome of Death | Safety Analysis Set |
| Listing 16.2.8.1 | Hematology and Coagulation Results and Change from Baseline | Safety Analysis Set |



| Listing 16.2.8.2 | Biochemistry Results and Change from Baseline | Safety Analysis Set |
|---|---|---|
| Listing 16.2.8.3 | Urinalysis Results and Change from Baseline | Safety Analysis Set |
| Listing 16.2.8.4 | Pregnancy Test Results (Females of Childbearing Potential only) | Safety Analysis Set |
| Listing 16.8.5 | Urine Drug Screen | Safety Analysis Set |
| Listing 16.2.9 | Vital Signs | Safety Analysis Set |
| Listing 16.2.10.1 | Electrocardiogram Results Part 1 | Safety Analysis Set |
| Listing 16.2.10.2 | Electrocardiogram Results Part 2 | Safety Analysis Set |
| Listing 16.2.11.1 | Physical Examinations | Safety Analysis Set |
| Listings 16.2.11.2 | Neurological Examination | Safety Analysis Set |
| Listing 16.2.12 | Columbia–Suicide Severity Rating Scale (C-SSRS) | Safety Analysis Set |
| Listing 16.2.13 | Electroencephalogram (EEG) Monitoring Test | Safety Analysis Set |
| Listing 16.2.14 | Magnetic Resonance Imaging (MRI) Test | Safety Analysis Set |
| Listing 16.2.15 | Positron Emission Tomography (PET) Test | Safety Analysis Set |
| Listing 16.2.16 | Alzheimer Disease History | Safety Analysis Set |
























































